CLINICAL TRIAL: NCT06751238
Title: An Open-label, Multicenter Study to Evaluate Pharmacokinetics, Safety and Tolerability up to 6 Years of Intravenous Secukinumab Infusions in Pediatric Participants With Juvenile Psoriatic Arthritis
Brief Title: Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability up to 6 Years of Intravenous (i.v.) Secukinumab in Pediatric Participants With Juvenile Psoriatic Arthritis (JPsA).
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457G22101
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Psoriatic Arthritis
Keywords: Pediatric; JPsA; Pharmacokinetic (PK); safety; Intravenous (i.v.); Secukinumab
MeSH Terms: conditions — Arthritis, Juvenile | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): Secukinumab administered intravenously in pediatric participants with JPsA
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — Intravenous secukinumab
  Other Names: AIN457

SUMMARY:
The purpose of this study is to determine the PK, safety and tolerability of multiple doses of intravenous (i.v.) secukinumab in pediatric participants with JPsA

DETAILED DESCRIPTION:
This is a multicenter, open-label study with an optional treatment extension period to evaluate pharmacokinetics, safety and tolerability (up to 6 years) of i.v. secukinumab in pediatric patients with JPsA.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants parent's or legal representative(s) written informed consent and child's assent, if appropriate, must be obtained before any study related activity or assessment is performed. Of note, if the participant reaches age of consent (as per local law) during the study, they will also need to sign the corresponding study ICF (Informed Consent Form).
* Males and females ≥2 years old to <18 years old at the time of screening.
* Confirmed diagnosis of JPsA according to the modified International League of Associations for Rheumatology (ILAR) classification criteria that must have occurred at least 6 months prior to screening.
* Active JPsA disease defined as ≥3 active joints (swollen or if not swollen must be both tender and limited range of motion) at baseline (BSL).
* Inadequate response (≥1 month) or intolerance to ≥1 Non-Steroidal Anti-Inflammatory Drug (NSAID) at screening.
* Inadequate response (≥2 months) or intolerance to ≥ 1 Disease Modifying Anti-Rheumatic Drug (DMARD) at screening.
* Concomitant use of the following second-line agents such as disease-modifying and/or immunosuppressive drugs to treat the JPsA will be allowed:

  * Stable dose of methotrexate (MTX) (maximum of 20 mg/ m2 BSA/ week) for at least 4 weeks prior to the BSL visit, with folic/folinic acid supplementation (according to standard medical practice of the center).
  * Stable dose of an oral corticosteroid (CS) at a prednisone equivalent dose of <0.2 mg/kg/day or up to 10 mg/day maximum, whichever is less, for at least 7 days prior to BSL.
  * Stable dose of no more than one NSAID for at least 1 week prior to BSL.

Key Exclusion Criteria:

* Participants with body weight less than 10 kg at screening.
* Use of other investigational drugs within 4 weeks or 5 half-lives of BSL, or until the expected pharmacodynamic effect has returned to BSL, whichever is longer.
* History of hypersensitivity to study drug or its excipients or to drugs of similar chemical classes.
* Participants with active inflammatory bowel disease or active uveitis at screening or BSL.
* Fulfilling diagnostic criteria for any International League of Associations for Rheumatology (ILAR ) juvenile idiopathic arthritis (JIA) category other than JPsA at BSL.
* Participants treated with prohibited medication
* Participants taking any non-biologic DMARD at screening except for MTX.
* Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Other inclusion/exclusion criteria may apply

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration on Day 1 | Pre-infusion and end of infusion (EOI) at Day 1
  Maximum concentration of secukinumab on Day 1
Maximum concentration at steady-state (Cmax, ss) | Preinfusion and EOI on Day 1, Day 29 and Day 57; weekly on Day 64, Day 71, Day 78, and Day 85; on Day 141 (pre-infusion if participant continues to the optional extension treatment or anytime during the visit if does not continue); preinfusion on Day 365
  Maximum concentration at steady-state.
Minimum concentration at steady-state (Cmin, ss) | Preinfusion and EOI on Day 1, Day 29 and Day 57; weekly on Day 64, Day 71, Day 78, and Day 85; on Day 141 (pre-infusion if participant continues to the optional extension treatment or anytime during the visit if does not continue); preinfusion on Day 365
  Minimum concentration at steady-state
Area under the concentration-time curve at steady-state (AUCtau, ss) | Preinfusion and EOI on Day 1, Day 29 and Day 57; weekly on Day 64, Day 71, Day 78, and Day 85; on Day 141 (pre-infusion if participant continues to the optional extension treatment or anytime during the visit if does not continue); preinfusion on Day 365
  Area under the concentration-time curve at steady-state during a dosing interval
Average concentration at steady-state (Cavg,ss) | Preinfusion and EOI on Day 1, Day 29 and Day 57; weekly on Day 64, Day 71, Day 78, and Day 85; on Day 141 (pre-infusion if participant continues to the optional extension treatment or anytime during the visit if does not continue); preinfusion on Day 365
  Average concentration at steady-state

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 20
  Number of participants with AEs and SAEs as a measure of safety and tolerability
Number of participants with clinically significant changes in clinical laboratory measures and vital signs. | Up to Week 20
  Number of participants with clinically significant changes in clinical laboratory measures and vital signs as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Florida, Gainesville, Florida
  - Ann and Robert H Lurie Childs Hosp, Chicago, Illinois
  - Levine Childrens Hospital, Charlotte, North Carolina
  - Univ Hosp Cleveland Medical Center, Cleveland, Ohio
  - Legacy Emanuel Research Hosp Portland, Portland, Oregon
  - Texas Arthritis Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com